CLINICAL TRIAL: NCT06265038
Title: A Prospective, Single Center, Confirmatory Investigation to Evaluate the Performance and Safety of ReSpace TiCell Cage Implants in Transforaminal Lumbar Interbody Fusion
Brief Title: Confirmatory Investigation to Evaluate the Performance and Safety of ReSpace TiCell Cage Implants in TLIF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sanatmetal Orthopaedic and Traumatologic Equipment Manufacturer Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SANAT-CAGE-2022
Record Dates: First submitted 2024-02-09; First posted 2024-02-20 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Degenerative Instability; Spondylolisthesis; Post-discectomy Syndrome; Post-traumatic Instability
Keywords: lumbar spinal; interbody fusion; interbody cage; 3D printing
MeSH Terms: conditions — Spondylolisthesis

STUDY DESIGN:
Intervention Model Description: Prospective, single-arm, open-label clinical trial. This clinical investigation addresses to collect data on clinical performance, effectiveness and safety of Sanatmetál's ReSpace TiCell Cage in human subjects following the good clinical practice according to the Medical Device Regulation (MDR) & EN ISO 14155:2020. The study is conducted in Hungary at National Center for Spinal Disorders.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prospective, single-arm, open-label clinical trial. (Other): Single center, prospective cohort, single-arm, open-label clinical trial Standard-of-care & Sanatmetal ReSpace TiCell Cage implantation A single-center study is sufficient to provide confirmatory data on performance and safety of the investigational device.
  Interventions: Device: ReSpace TiCell Cage

INTERVENTIONS:
Device: ReSpace TiCell Cage — ReSpace TiCell Cages are anatomically shaped interbody spacer implants with curved contour. These implants intended to be inserted into the intervertebral disc space for intervertebral body fusion. The interbody spacers are designed to restore height and lordotic angle in the spine. The spacers have teeth on the endplate-engaging surfaces to provide stability, resist shear and rotational forces, and to help prevent migration of the spacer within the disc space. The open central cavity on them allows for placement of graft material allowing for subsequent bone growth through the interior of the devices.
  ReSpace TiCell Cages are indicated for lumbar spine stabilization (between L.I.-S.I. segments). TLIF spine surgery will be combined with posterior fixation using pedicle screws and rods.

SUMMARY:
The primary objective of this study is to confirm superiority for the efficacy of the ReSpace Ticell Cage implants in Transforaminal Lumbar Interbody Fusion compared to state-of-the-art.

The secondary objective of the study is to evaluate further efficacy and safety of the ReSpace Ticell Cage implants in Transforaminal Lumbar Interbody Fusion with the following secondary efficacy and safety objectives:

* To evaluate if implantation causes significant reduction in patient's back, hip/buttock, and leg pain.
* To evaluate if implantation causes significant increase quality of life of the patients.
* To evaluate if using the device can be considered as safe overall.

DETAILED DESCRIPTION:
Degenerative disc and facet joint disease of the lumbar spine is common in the ageing population and is one of the most frequent causes of disability. Lumbar spondylosis may result in mechanical back pain, radicular and claudicant symptoms, reduced mobility and poor quality of life. Surgical interbody fusion of degenerative levels is an effective treatment option to stabilize the painful motion segment, and may provide indirect decompression of the neural elements, restore lordosis and correct deformity. Lumbar interbody fusion (LIF) involves placement of an implant (cage, spacer or structural graft) within the intervertebral space after discectomy and endplate preparation. At this time LIF is performed using five main approaches; posterior lumbar interbody fusion (PLIF), transforaminal lumbar interbody fusion (TLIF), oblique lumbar interbody fusion/anterior to psoas (OLIF/ATP), anterior lumbar interbody fusion (ALIF) and lateral lumbar interbody fusion (LLIF). There is no clear definitive evidence for one approach being superior to another in terms of fusion or clinical outcomes. These operations can also be performed using mini-open or minimally invasive (MIS) approaches, however it has not yet been demonstrated that MIS-TLIF is clinically superior to traditional open TLIF procedure. Interbody fusion is preferable to postero-lateral 'onlay' fusion techniques due to lower rates of postoperative complications and pseudoarthrosis.

Posterior interbody fusion (PLIF), combined with segmental instrumentation, has become increasingly popular since it was first described by Mercer in 1936 and expanded upon by Cloward. More recently however, the transforaminal approach to the intervertebral disc, known as transforaminal lumbar interbody fusion (TLIF), has gained popularity. Originally described by Harms in the late 1990s, the TLIF has arguably developed into the most commonly performed and efficacious posterior interbody fusion method in modern spine surgery.

Transforaminal lumbar interbody fusion (TLIF) utilizes a more lateral window in order to access the interbody space without excessive dural retraction. Theoretical advantages of TLIF include increased fusion success, more complete foraminal decompression, better correction of deformity, and more effective treatment of discogenic pain.

Transforaminal lumbar interbody fusion (TLIF) have demonstrated excellent fusion rates with acceptable complication profiles for treating single and multilevel lumbar disc pathology and instability. TLIF have been shown to be superior to posterolateral fusion alone for deformity correction and more cost effective than anterior interbody combined with posterior segmental instrumentation.

ELIGIBILITY:
Inclusion Criteria:

Each subject must meet all the following criteria to be enrolled in this study:

All subjects who had previously indicated for TLIF surgery can participate in this study, with the following evidence:

1. Has degenerative disease of the lumbosacral spine in one or two adjacent levels (L1 to S1), manifested by:

   1. Low back pain, or
   2. Irradiating leg or buttock pain, paresthesia, numbness, or weakness, or
   3. History of neurogenic claudication.
2. Has radiographic evidence (e.g. CT, MRI, x-ray, etc.) of degenerative lumbosacral disease including at least one of the following:

   1. Instability as defined by ≥3 mm translation or ≥5-degree angulation
   2. Decreased disc height, on average by ≥2 mm, but dependent upon the spinal level
   3. Scarring/thickening of ligamentum flavum or annulus fibrosis
   4. Herniated nucleus pulposus
   5. Vacuum phenomenon
   6. Grade 1 spondylolisthesis/retrolisthesis based on the Meyerding classification (Meyerding, Henry William, 1932), or lateral listhesis demonstrated by coronal plane translation (slippage) of the superior (cranial) vertebral body lateral to the inferior (caudal) vertebral body less than or equal to 3mm, or
   7. Stenosis, or narrowing, of the lumbar spinal canal and/or intervertebral foramen requiring significant decompression leading to segmental instability, or
   8. Recurrent disc herniation

Further inclusion criteria:

* Skeletally mature adults ages 18 - 80 years of age
* Able to read and understand all documents used in this study, including the informed consent and patient-reported outcome questionnaires

Exclusion Criteria:

Subjects meeting any of the following criteria will be excluded from the study:

1. Prior surgical procedure at the involved or adjacent spinal levels (e.g. stabilization, fusion, arthroplasty and/or other non-fusion procedures). Prior microdiscectomy, discectomy, laminectomy, decompression surgery at the target or adjacent levels is allowed.
2. Significant lumbar instability defined as sagittal listhesis greater than Grade 2 at any involved level using the Meyerding Classification or lateral listhesis greater than 3 mm at any involved level.
3. Planned use of an internal or external bone growth stimulator.
4. Lumbar scoliosis >30 degrees.
5. Patients who had a previous diagnosis of osteoporosis with a Tscore of -2.5 or below in the last 12 months. If subject has a prevalent fragility fracture and a T-score hasn't been assessed in the last 12 months, a DEXA (dual x-ray absorptiometry) scan will need to be obtained.
6. Morbidly obese, as defined by a Body Mass Index (BMI) >40.
7. Presence of active malignancy or prior history of malignancy (noninvasive basal cell carcinoma of the skin and non-invasive squamous cell carcinoma localized only to the skin is allowed).
8. Overt or active bacterial infection, either local to surgical space or systemic.
9. Has undergone administration of any type of corticosteroid, antineoplastic, immunostimulant, or immunosuppressive agents, or medications known to inhibit with the healing of bone or soft tissue within 30 days prior to implantation of the assigned treatment

   1. This includes patients ≥ 65 years of age taking warfarin with documented diagnosed osteoporosis. All other patients taking warfarin should washout for at least 5 days prior to treatment
   2. Use of steroidal inhalers, short-term NSAID use, and shortterm steroidal use (e.g. Medrol Dosepak) is allowed pre and postoperatively. For this clinical study, short-term use is defined as ≤ two weeks.
   3. Use of NSAIDs and/or steroids for longer than two weeks postoperatively through the 24 Month Follow-Up Visit is not recommended. Such patients must be excluded from data analysis in case of non-fusion.
10. Co-morbidities, which in the investigator's opinion, precludes the subject from being a surgical candidate.
11. Autoimmune disease, which in the investigator's opinion, is known to affect bone metabolism or the spine (e.g., spondyloarthropathies, juvenile arthritis, rheumatoid arthritis, Graves' disease, Hashimoto's thyroiditis).
12. Any endocrine or metabolic disorder, which in the investigator's opinion, is known to affect osteogenesis (e.g., Paget's disease, renal osteodystrophy, Ehlers-Danlos syndrome, or osteogenesis imperfecta).
13. Known hypersensitivity or allergy to any components of the study treatments including, but not limited to bone morphogenetic proteins (BMPs); injectable collagen; protein pharmaceuticals (e.g.: monoclonal antibodies or gamma globulins); bovine collagen products; and/or instrumentation materials (e.g., titanium, titanium alloy, cobalt chrome, cobalt chrome alloy, or PEEK).
14. History of any allergy resulting in anaphylaxis.
15. Is mentally incompetent. If questionable, obtain psychiatric consult.
16. Treatment with an investigational therapy (drug, device, and/or biologic) targeting spinal conditions within 3 months prior to implantation surgery, treatment with any other investigational therapies within 30 days prior to implantation surgery, or such treatment is planned during the 24-month period following implantation of the study treatment.
17. Pregnancy and breastfeeding.
18. A documented diagnosis of substance use disorder (Nicotine use is allowed.)
19. Any condition, which in the investigator's opinion, would interfere with the subject's ability to comply with study instructions, which might confound data interpretation.
20. Subject is considered to belong to a vulnerable population.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
CT imaging_1 - cumulative fusion rate | At visit 4 (Month 24)
  For the determination of the cumulative fusion rate, radiographic evaluation (CT imaging with fine-cut axial and multiplanar reconstruction views) will be conducted by 2 independent examiners.
CT imaging_2 - fusion status | At visit 4 (Month 24)
  Standing flexion-extension angle will be measured with dynamic plain radiography to evaluate mobility to determine the fusion status.

SECONDARY OUTCOMES:
Visual Analog Scale | At visits 1/2/3/4 (Months 3/6/12 and 24)
  The severity of back, hip/buttock, and leg pain will each be evaluated in all study subjects using a 100-mm Visual Analog Scale (VAS). Minimum value is 0mm, maximum value is 100mm. The low value means low intensity of the pain, which is the aim of the treatment.
Oswestry Disability Index (ODI) | At visits 1/2/3/4 (Months 3/6/12 and 24)
  Oswestry Disability Index (ODI) is a validated, independent outcome measure. It is one of the principal condition-specific outcome measures used in the management of spinal disorders and in patients with low back pain. The questionnaire contains 10 questions. There are 6 possible answers available to each questions. The 1. answer means each time the lowest pain, which is the aim of the treatment. At the end the doctor calculate a rate of the patient pain in %.

OTHER OUTCOMES:
AE and ADE | During the study (32 months)
  To prove the safe and effective use of the medical device. Number of patients with Adverse Events (AE) and Adverse Device Effects (ADE) are administered and observed during the study.
Complications | During the study (32 months)
  To prove the safe and effective use of the medical device. The rate of complications is administered and observed during the study.
Surgical revisions | During the study (32 months)
  To prove the safe and effective use of the medical device. The rate of surgical revisions is administered and observed during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Aron Lazary, MD, PhD, Principal Investigator — National Center for Spinal Disorders
Locations (1):
- National Center for Spinal Disorders, Budapest, Pest County, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ajiboye RM, Alas H, Mosich GM, Sharma A, Pourtaheri S. Radiographic and Clinical Outcomes of Anterior and Transforaminal Lumbar Interbody Fusions: A Systematic Review and Meta-analysis of Comparative Studies. Clin Spine Surg. 2018 May;31(4):E230-E238. doi: 10.1097/BSD.0000000000000549. PMID 28622187
- [Result] Kim JS, Kang BU, Lee SH, Jung B, Choi YG, Jeon SH, Lee HY. Mini-transforaminal lumbar interbody fusion versus anterior lumbar interbody fusion augmented by percutaneous pedicle screw fixation: a comparison of surgical outcomes in adult low-grade isthmic spondylolisthesis. J Spinal Disord Tech. 2009 Apr;22(2):114-21. doi: 10.1097/BSD.0b013e318169bff5. PMID 19342933
- [Result] Kim JS, Lee KY, Lee SH, Lee HY. Which lumbar interbody fusion technique is better in terms of level for the treatment of unstable isthmic spondylolisthesis? J Neurosurg Spine. 2010 Feb;12(2):171-7. doi: 10.3171/2009.9.SPINE09272. PMID 20121352
- [Result] Crandall DG, Revella J. Transforaminal lumbar interbody fusion versus anterior lumbar interbody fusion as an adjunct to posterior instrumented correction of degenerative lumbar scoliosis: three year clinical and radiographic outcomes. Spine (Phila Pa 1976). 2009 Sep 15;34(20):2126-33. doi: 10.1097/BRS.0b013e3181b612db. PMID 19752698
- [Result] Dorward IG, Lenke LG, Bridwell KH, O'Leary PT, Stoker GE, Pahys JM, Kang MM, Sides BA, Koester LA. Transforaminal versus anterior lumbar interbody fusion in long deformity constructs: a matched cohort analysis. Spine (Phila Pa 1976). 2013 May 20;38(12):E755-62. doi: 10.1097/BRS.0b013e31828d6ca3. PMID 23442780
- [Result] Faundez AA, Schwender JD, Safriel Y, Gilbert TJ, Mehbod AA, Denis F, Transfeldt EE, Wroblewski JM. Clinical and radiological outcome of anterior-posterior fusion versus transforaminal lumbar interbody fusion for symptomatic disc degeneration: a retrospective comparative study of 133 patients. Eur Spine J. 2009 Feb;18(2):203-11. doi: 10.1007/s00586-008-0845-0. Epub 2009 Jan 6. PMID 19125304
- [Result] Hee HT, Castro FP Jr, Majd ME, Holt RT, Myers L. Anterior/posterior lumbar fusion versus transforaminal lumbar interbody fusion: analysis of complications and predictive factors. J Spinal Disord. 2001 Dec;14(6):533-40. doi: 10.1097/00002517-200112000-00013. PMID 11723406
- [Result] Levin JM, Tanenbaum JE, Steinmetz MP, Mroz TE, Overley SC. Posterolateral fusion (PLF) versus transforaminal lumbar interbody fusion (TLIF) for spondylolisthesis: a systematic review and meta-analysis. Spine J. 2018 Jun;18(6):1088-1098. doi: 10.1016/j.spinee.2018.01.028. Epub 2018 Feb 13. PMID 29452283
- [Result] Carreon LY, Glassman SD, Ghogawala Z, Mummaneni PV, McGirt MJ, Asher AL. Modeled cost-effectiveness of transforaminal lumbar interbody fusion compared with posterolateral fusion for spondylolisthesis using N(2)QOD data. J Neurosurg Spine. 2016 Jun;24(6):916-21. doi: 10.3171/2015.10.SPINE15917. Epub 2016 Feb 19. PMID 26895529
- [Result] Fujimori T, Le H, Schairer WW, Berven SH, Qamirani E, Hu SS. Does Transforaminal Lumbar Interbody Fusion Have Advantages over Posterolateral Lumbar Fusion for Degenerative Spondylolisthesis? Global Spine J. 2015 Apr;5(2):102-9. doi: 10.1055/s-0034-1396432. Epub 2014 Dec 1. PMID 25844282
- [Result] Ghasemi AA. Transforaminal lumbar interbody fusion versus instrumented posterolateral fusion In degenerative spondylolisthesis: An attempt to evaluate the superiority of one method over the other. Clin Neurol Neurosurg. 2016 Nov;150:1-5. doi: 10.1016/j.clineuro.2016.08.017. Epub 2016 Aug 21. PMID 27565009
- [Result] Owens RK 2nd, Carreon LY, Djurasovic M, Glassman SD. Relative benefit of TLIF versus PSF stratified by diagnostic indication. J Spinal Disord Tech. 2014 May;27(3):144-7. doi: 10.1097/BSD.0b013e3182867470. PMID 24945292
- [Result] Pooswamy S, Muralidharagopalan NR, Subbaiah S. Transforaminal lumbar interbody fusion versus instrumented posterolateral fusion in Grade I/II spondylolisthesis. Indian J Orthop. 2017 Mar-Apr;51(2):131-138. doi: 10.4103/0019-5413.201703. PMID 28400657
- [Result] Makanji H, Schoenfeld AJ, Bhalla A, Bono CM. Critical analysis of trends in lumbar fusion for degenerative disorders revisited: influence of technique on fusion rate and clinical outcomes. Eur Spine J. 2018 Aug;27(8):1868-1876. doi: 10.1007/s00586-018-5544-x. Epub 2018 Mar 15. PMID 29546538